CLINICAL TRIAL: NCT05580861
Title: Phase I/II Clinical Trial Assessing the Combination of Sulfasalazine With Standard of Care Induction Therapy in Newly Diagnosed Acute Myeloid Leukemias (AML) Patients 60 Years or Older- the SALMA Study
Brief Title: Sulfasalazine in AML Treated by Intensive Chemotherapy: Elderly Patients-first Line Treatment
Acronym: SALMA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP211176
Record Dates: First submitted 2022-09-26; First posted 2022-10-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sulfasalazine

STUDY DESIGN:
Intervention Model Description: Phase I dose-finding design unsing the continueal reassessment method, followed by a dose expansion cohort using a Simon's phase II design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort : Patients with acute myeloid leukemia (Experimental)
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — Sulfazalazine 500mg-tablets ; 7 dose levels explored in the phase I part of the trial.

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous clonal myeloid neoplasm where abnormal proliferation and impaired differentiation of hematopoietic stem and myeloid progenitor cells impedes normal hematopoiesis. Sulfasalazine (SSZ) is a broadly available, well tolerated anti-inflammatory medicine approved for the treatment of ulcerative colitis and rheumatoid arthritis. Intact SSZ, but not its metabolites 5-aminosalicylic acid and sulfapyridine, competitively inhibits xCT.21 SSZ is thus an ideal candidate for drug repurposing in AML.The purpose of this phase I study is to evaluate the safety and feasibility of such strategy, provide preliminary signals of efficacy, and identify potential biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or older
* With newly diagnosed acute myeloid leukemia (AML) (short course treatment with hydroxyurea and or steroids is acceptable). Patients with AML secondary to an antecedent Myelodysplastic Syndromes (MDS) or Myeloproliferative Neoplasms (MPN) are eligible, as those with therapy-related AML.
* Eligible for intensive chemotherapy in the investigator's opinion
* Leukaemia-associated immunophenotypes (LAIP) detected at screening allowing flow cytometry (FCM)-based Minimal Residual Disease monitoring (Phase II only).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Aspartate transaminase (AST) and Alanine transaminanse (ALT) ≤ 3.0 times upper the limit of normal (ULN) and total and direct serum bilirubin ≤ 1.5 x ULN unless considered due to leukemia Estimated glomerular filtration rate (GFR) ≥ 50 mL/min according to the MDRD equation
* Written informed consent obtained prior to any screening procedures
* Eligible for National Health Insurance in France

Exclusion Criteria:

* Myeloid Sarcoma with < 20% bone marrow blasts
* Patient who has received a vaccine injection with live-attenuated virus in the last three weeks
* Proven central nervous system leukemic involvement
* Favorable risk cytogenetics: t(15;17), t(8;21), inv(16) or t(16;16) or presence of PML-RARA, RUNX1-RUNX1T1 or CBFB-MYH11 fusion transcript.
* Presence of FLT3-ITD or TKD mandating treatment with midostaurin.
* Concurrent therapy with any cytotoxic drug within 3 weeks before the first study dose. Only hydroxyurea for the control of blood counts is permitted.
* Patients planned to received CPX-351 for myelodysplasia-related changes or therapy-related AML.

Previous treatment with sulfasalazine in the last 5 years or ongoing treatment with sulfasalazine or 5-aminosalicylic acid (5-ASA) for ulcerative colitis or inflammatory rheumatisms.

* History of allergy SSZ, one of its metabolites (5-aminosalicylic acid, 5-ASA) or mesalazine, other sulfonylarylamines sulfonamides or salicylates, or sulfasalazine excipients History of allergic reaction to idarubicin or idarubicin excipients
* History of allergic reaction to cytarabine or cytarabine excipients
* Known glucose 6-phosphate dehydrogenase deficiency.
* Known acute intermittent porphyria or porphyria variegata.
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate treatment).
* Other uncontrolled or active malignant disease within prior 12 months (excluding myelodysplastic syndrome; cutaneous basal cell carcinoma, "in-situ" carcinoma of the cervix or breast, or other local malignancy excised).
* Known human immunodeficiency virus (HIV) infection or HIV-related malignancy.
* Clinically active hepatitis B or hepatitis C infection.
* Inability to swallow. Known malabsorption syndrome or other condition that may significantly impair absorption of oral study medications.
* Participation in another therapeutic interventional clinical study within 30 days of enrolment.
* Administration of any therapy considered investigational (i.e., used for non-approved indications(s) or in the context of a research investigation) within 5 drug half-lives (whichever is longer) prior to the first dose of study drug.
* Previous treatment by anthracyclines
* Any contraindication to use anthracyclines including uncontrolled coronary disease, severe renal failure, severe hepatic failure, recent myocardial infarction, symptomatic congestive heart failure, severe cardiomyopathy, significant arrhythmia as estimated by the investigator or left-ventricule ejection fraction (LVEF) <53% as assessed by echocardiography or Multigated Acquisition Scan (MUGA), anterior treatment by idarubicin and/or anthracyclines and anthracènediones beyond the maximum cumulative dose.
* Any contraindication to use cytarabine including degenerative and toxic encephalopathy.
* Any condition requiring treatment with digoxin.
* Any of concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study.
* Females who are pregnant or breastfeeding.
* In a man whose sexual partner is a woman of childbearing potential, unwillingness or inability of the man or woman to use a highly effective contraceptive method for the entire treatment period and for at least 6 months after completion of protocol treatment.

Highly effective contraception methods include: combined (estrogen and progestogen containing) hormonal methods associated with inhibition of ovulation, intra-uterine device; surgical sterilization (including bilateral tubal occlusion, partner's vasectomy) or sexual abstinence if this is the preferred and usual lifestyle of the patient.

Male patients must not freeze or donate sperm starting at screening and throughout the treatment period and 3 months after the administration of the final dose of study medication.

- In a heterosexually active woman of childbearing potential, unwillingness or inability to use a highly effective contraceptive method (as described above) for the entire treatment period and for at least 6 months after the administration of the final dose of study medication.

Women are not regarded as of childbearing potential if they are post-menopausal (at least 2 years without menses) or are surgically sterile (at least 1 month before enrollment).

Female patients must not donate or retrieve, for their own use, ova from the time of screening and throughout the treatment period, and for 12 weeks after the administration of the final dose of study medication.

Female patients must agree not to breastfeed from the time of screening and throughout the protocol period, and for (5 half-lives) days after the administration of the final dose of study medication.

Adults subjects to a legal protection order or unable to give their consent

- Persons deprived of their freedom by judicial or administrative decision, person hospitalized without their consent by virtues of French Public Health Code articles L 3212-1 and L3213-1 and who are not subject to the provisions of article L 1121-8.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (for phase I part of the trial) | 42 days
  Defined as any of the following events:
  * Prolonged myelosuppression defined as Grade ≥ 3 Neutropenia or Thrombocytopenia on Day 42 from start of therapy or later without evidence of leukemia (assessed by bone marrow aspiration and/or biopsy)
  * Grade ≥3 hemorrhages until day 42.
  * Grade ≥3 non- hematological toxicity until day 42 with the exception of: Grade 3 infection, grade 3 fever with neutropenia (NB. grade 4 infections and grade 4 fever with neutropenia are considered as DLTs), Grade ≥3 nausea, vomiting or diarrhea that can be managed to ≤ Grade 2 within 72 hours of symptomatic treatment, Grade ≥3 asymptomatic liver enzymes elevation that improves to ≤ Grade 2 within 72 hours of onset, Grade ≥3 tumor lysis syndrome that resolves within 72 hours of onset with medical treatment
Minimal Residual Disease (MRD)-negative Complete Response (for phase II part of the trial) | Day 28 to 42
  Defined as:
  * Complete Remission CR or CRi (CR with incomplete hematologic recovery, meaning CR with platelet count <100,000/μL or absolute neutrophil count <1000/μL) and CRh (CR with partial hematologic recovery, meaning CR not fulfilling CR or CRi peripheral blood count criteria but with platelet count >50,000/μL AND absolute neutrophil count >500/μL).
  * MRD-negativity is defined as an 8-color bone marrow FCM MRD < 0.1% at EOI.
  * Of note, NPM1 (nucleoplasmin)-transcript based MRD in the Bone Marrow and Peripheral Blood will be carried as exploratory endpoint in NPM1-mutated patients.

SECONDARY OUTCOMES:
Adverse events | Month 12
  Adverse events (AE), treatment emergent adverse events (TEAE) and treatment-related TEAEs will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Peak plasma concentration (Cmax) of Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of Peak Plasma Concentration (Cmax), in the phase I part of the study
Time of peak plasma concentration (Tmax) of Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of Time of peak plasma concentration (Tmax) of Sulfazalazine, in the phase I part of the study
Area under the plasma concentration versus time curve (AUC) for Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of area under the plasma concentration versus time curve (AUC), in the phase I part of the study
Clearance (Cl) of Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of clearance (Cl), in the phase I part of the study
Mean residence time (MRT) of Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of mean residence time (MRT), in the phase I part of the study
Distribution volume (Vd/F) of Sulfazalazine | Day 1, 4 and 15
  Pharmacokinetics of Sulfazalazine in terms of distribution volume (Vd/F), in the phase I part of the study
Plasma levels of malondialdehyde | Day 1, 2
  Pharmacodynamics with plasma levels of malondialdehyde (MDA)
Plasma levels of glutathione | Day 1, 2
  Pharmacodynamics with plasma levels of glutathione (reduced/oxidized)
Reactive Oxygen Species (ROS) levels of peripheral blood mononuclear cells | Day 1, 2
  In patients with circulating leukemic cells, ROS levels of peripheral blood mononuclear cells by flow cytometry
Response | End of induction treatment - day 28 to 42
  Response at end of induction assessment (day 28-42) as per European LeukemiaNet (ELN) Criteria.
Nucleophosmin (NPM1)-transcript based Minimal Residual Disease (MRD) | End of induction treatment - day 28 to 42
  NPM1-transcript based MRD in the bone marrow and peripheral blood in NPM1-mutated patients
Next-generation sequencing (NGS)-based Minimal Residual Disease (MRD) | End of induction treatment - day 28 to 42
  NGS-based MRD in all patients
Event-free survival | 12 months
  Event-free survival (EFS) defined as the time between inclusion and the first of the following events:
  * Non achievement of hematologic response (including complete response (CR), CR with incomplete hematologic recovery (CRi), CR with partial hematologic recovery (CRh))
  * Hematologic relapse or progressive disease
  * Initiation of any subsequent anti-leukemic therapy (excluding hydroxyurea)
  * Death
Duration of response (DOR) | 12 months
  Duration of response (DOR)
Relapse-free survival | 12 months
  Relapse-free survival (RFS) defined as the time between inclusion and the first of the following events:
  * Hematologic relapse or progressive disease
  * Death
Overall survival | 12 months
  Overall survival (OS), defined as the time between inclusion and death
Incidence of subsequent allogeneic hematopoietic stem cell transplant | 12 months
  Incidence of subsequent allogeneic hematopoietic stem cell transplant (HSCT), overall and in responding patients specifically
Targeted gene sequencing | Inclusion and end of induction (day 28 to 42)
  Targeted sequencing of a panel of genes recurrently mutated in AML, on bone marrow and peripheral blood samples
SLC7A11 expression | Inclusion and end of induction (day 28 to 42)
  SLC7A11 expression by flow cytometry (FCM) and/or western blot (WB), on bone marrow and peripheral blood samples
Genotyping of ABCG2 rs2231142 polymorphisms | Inclusion and end of induction (day 28 to 42)
  Genotyping of ABCG2 rs2231142 polymorphisms, on bone marrow and peripheral blood samples, in consenting patients
NAT2 genotype | Inclusion and end of induction (day 28 to 42)
  NAT2 genotype (NAT2*4, NAT2*5B, NAT2*6A, NAT2*7B), in consenting patients
RNA-based antioxidogram | Inclusion and end of induction (day 28 to 42)
  RNA-based expression patterns of major enzymes involved in the antioxidant cellular response (as described in Picou et al, Blood Advances 2019)
Antioxidant score | Inclusion and end of induction (day 28 to 42)
  Antioxidant score is a summary measure of expression patterns of major enzymes involved in the antioxidant cellular response (as described in Picou et al, Blood Advances 2019)
Expression of NRF2 target genes | Inclusion and end of induction (day 28 to 42)
  Expression of NRF2 target genes (NRF2 score) on bone marrow samples

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Amiens, Amiens
  - Hôpital Avicenne, Bobigny
  - CHU Caen, Caen
  - CHU Henri Mondor, Créteil
  - Centre Hospitalier Lyon Sud, Lyon, Lyon
  - Hôpital de la Conception, AP-HM, Marseille
  - CHU Nice, Nice
  - AP-HP Hôpital Saint Louis, Paris
  - AP-HP Hôpital Cochin, Paris
  - Centre Henri Becquerel, Rouen
  - CHU Tours, Tours
  - CH Mignot, Versailles
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided